CLINICAL TRIAL: NCT03679195
Title: Impact of a Supplementation With Grape Seed and Cranberry Extracts on Ambulatory Blood Pressure
Brief Title: Effect of Polyphenols Combined to L-citrulline on Ambulatory Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Atrium Innovations (Industry)
Responsible Party: Principal Investigator, Benoit Lamarche, PhD, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INAF_NO_2017-207
Record Dates: First submitted 2018-09-14; First posted 2018-09-20 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
Keywords: 24h ambulatory blood pressure vascular function inflammation
MeSH Terms: conditions — Hypertension | interventions — Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NO Ultra (Nitric Oxid Ultra Capsules) (Experimental): 764 mg/day of cranberry and grape seed extracts (containing polyphenols) and 2 g/day of L-citrulline. Participants will have to take daily 2 NO Ultra capsules (containing 382 mg cranberry and grape seed extracts / 1 g L-citrulline) between breakfast and lunch and 2 other NO Ultra capsules between lunch and dinner.
  Interventions: Dietary Supplement: NO Ultra
- Placebo (Cellulose Capsules) (Placebo Comparator): Participants will consume cellulose capsules that are similar in shape and size to the NO ultra product, i.e. 2 capsules between breakfast and lunch and 2 other capsules between lunch and dinner.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NO Ultra — 6-week supplementation period with 764 mg/day of cranberry and grape seed extracts (containing polyphenols) and 2 g/day of L-citrulline Participants will have to take daily 2 NO Ultra capsules (containing 382 mg cranberry and grape seed extracts / 1 g L-citrulline) between breakfast and lunch and 2 other NO Ultra capsules between lunch and dinner.
  Arms: NO Ultra (Nitric Oxid Ultra Capsules)
Dietary Supplement: Placebo — 6-week supplementation period with placebo capsules (the active ingredients will be replaced by cellulose)
  Participants will have to take 2 capsules of cellulose between breakfast and lunch and 2 capsules between lunch and dinner to match the number of capsules ingested daily by the NO Ultra group.
  Other Names: Cellulose capsules
  Arms: Placebo (Cellulose Capsules)

SUMMARY:
The general objective of this project is to investigate the chronic effect of consuming supplements combining polyphenols from cranberry and grape seed extracts and L-citrulline (Nitric Oxide Ultra capsules, Pure Encapsulations, Sudbury, MA) on 24-hour ambulatory blood pressure, markers of vascular function and plasma biomarkers of inflammation in adults with pre-hypertension.

The study will be undertaken according to a double-blind, parallel, randomized, placebo controlled design and will be conducted at the Institute of Nutrition and Functional Foods (INAF) of Laval University. The study will involve a total of 73 adult men and women. Included subjects will be randomly assigned to a 6-week period of supplementation with Nitric Oxide (NO) Ultra capsules or placebo (cellulose capsules). The outcomes are the chronic changes after supplementation with NO Ultra capsules compared with the placebo in: 24-hour ambulatory diastolic and systolic blood pressure, levels of blood lipids and inflammation markers, levels of blood and cutaneous markers of vascular function.

DETAILED DESCRIPTION:
There is now evidence that blood pressure, vascular function and inflammation are intimately associated with cardiovascular disease. It is also clear that several dietary components including polyphenols and L-citrulline can modify blood pressure control. However, based on the studies available so far, it is difficult to draw firm conclusion on the potential impact of a dietary supplement combining polyphenols and L-citrulline on ambulatory blood pressure in pre-hypertensive subjects at risk to develop hypertension and cardiovascular disease. To the best of our knowledge, no study has yet investigated the chronic impact of combined polyphenols and L-citrulline on both ambulatory blood pressure and vascular function/inflammation.

The present supplementation based on polyphenols and L-citrulline may represent for pre-hypertensive subjects a new dietary modality to manage blood pressure as part of healthy eating.

The study will be undertaken according to a double-blind, parallel, randomized, placebo controlled design and will be conducted at the Institute of Nutrition and Functional Foods (INAF) of Laval University. A total of 73 adult men and women will be recruited based primarily on blood pressure criteria in the Quebec City metropolitan area. Participants will be randomly assigned to a 6-week period of supplementation with Nitric Oxide Ultra capsules or placebo (cellulose capsules). Participants in the NO Ultra group will be supplemented with 764 mg/day of cranberry and grape seed extracts (containing polyphenols) and 2 g/day of L-citrulline. Participants will have to take daily 2 capsules (NO Ultra or placebo) between breakfast and lunch and 2 capsules (NO Ultra or placebo) between lunch and dinner. Specifically, capsules will be taken with water and no foods, and at least one-hour apart meals. Office and 24-hour ambulatory blood pressure, blood lipids, cutaneous and plasma markers of vascular function, plasma inflammation biomarkers and anthropometric characteristics will be measured at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18-75 years
* For women with child-bearing potential, acceptable effective contraceptive methods are: total abstinence, hormonal birth control methods (oral, injectable, transdermal or intra-vaginal), intrauterine devices, confirmed successful vasectomy of partner
* Stable weight for at least three 3 months (±5lbs)
* Mean daytime SBP between 125 and 134.9 mmHg and DBP < 85 mmHg
* Otherwise healthy individuals

Exclusion Criteria:

* Women during a peri-menopausal period
* Pregnant/breastfeeding women
* Mean daytime SBP <125 or >134.9 mmHg or DBP ≥85 mmHg
* History of cardiovascular disease, type 2 diabetes, monogenic dyslipidemia or endocrine disorders
* Use of anticoagulants or thrombocyte aggregation inhibitors, chemotherapeutic agents, anti-inflammatory drugs, medication for blood lipids, diabetes, hypertension, erectile dysfunction or auto-immune diseases
* Any clinical signs or laboratory evidence for inflammatory, gastrointestinal, endocrine, renal, pulmonary, neurological, cardiovascular, metabolic, haematological problem or cancer
* Kidney stones
* Excess alcohol consumption (> 14 consumptions/week) or drug consumption
* Hypersensitivity/allergy to one of the ingredients (including non-medicinal ingredients) in NO Ultra supplement/placebo
* Use of additional cranberry/grape seed extract or citrulline products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory diastolic blood pressure | 6 weeks (end-point value)
  Comparison of the change from baseline in 24-hr ambulatory diastolic blood pressure at 6-wk between the NO Ultra group and the placebo group.

SECONDARY OUTCOMES:
24-hour ambulatory systolic blood pressure | 6 weeks (end-point value)
  Comparison of the change from baseline in 24-hr ambulatory systolic blood pressure at 6-wk between the NO Ultra group and the placebo group.
Blood Lipids | 6 weeks (end-point value)
  Comparison of the change from baseline in serum total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, non HDL cholesterol, TG, and apolipoprotein B levels as well as in the total cholesterol/HDL cholesterol ratio at 6-wk between the NO Ultra group and the placebo group.
  The concentration of the above lipids will be assessed on a Roche/Hitachi Modular analytical system (Roche Diagnostics) according to the manufacturer's specifications and using proprietary reagents. Serum LDL cholesterol concentrations will be calculated using the Friedewald equation.
Vascular function | 6 weeks (end-point value)
  Comparison of the change from baseline in serum markers of vascular function including concentrations of angiotensin-converting enzyme (ACE), angiotensin-II (A-II), aldosterone (ALDOS), soluble forms of intercellular adhesion molecules (sICAM-1), soluble form of vascular cell adhesion molecule-1 (sVCAM-1) and soluble form of E-selectin (sE-selectin), as well as in the skin concentration of advanced glycation end products (AGEs) at 6-wk between the NO Ultra group and the placebo group.
  Plasma concentrations of ACE, A-II, aldosterone ALDOS, sICAM-1, sVCAM-1 and sE-selectin will be determined using commercial ELISA kits for the human form of these markers. Measurement of the skin concentration of AGEs iwill be performed using a sensitive optical measurement device called AGE scanner (DiagnOptics, Groningen, The Netherlands).
Inflammation biomarkers | 6 weeks (end-point value)
  Comparison of the change from baseline in serum levels of C-reactive protein (CRP), interleukin-6 (IL-6), IL-18 and tumor necrosis factor alpha (TNF-a) at 6-wk between the NO Ultra group and the placebo group.
  Serum CRP concentrations will be measured using of the Behring Latex-Enhanced highly sensitive assay on the Behring Nephelometer BN-100 system. Serum IL-6, IL-18, and TNF-alpha concentrations will be determined using commercial ELISA kits for the human form of these cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Funtional Foods, Québec, Canada